CLINICAL TRIAL: NCT02002702
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Assess the Safety, Tolerability and Pharmacokinetics of Serelaxin When Added to Standard Therapy in Japanese Acute Heart Failure Patients
Brief Title: Study of Safety, Tolerability and Pharmacokinetics of Serelaxin in Japanese Acute Heart Failure (AHF) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRLX030A1201
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure (AHF),; Japanese,; Safety and tolerability, Pharmacokinetics,; Renal Impairment
MeSH Terms: conditions — Hemophilia A; Renal Insufficiency | interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Serelaxin 10 mcg/kg/Day (Experimental): Participants received 10 mcg/kg/day serelaxin as continuous i.v. infusion for 48 hours.
  Interventions: Drug: Serelaxin
- Serelaxin 30 mcg/kg/Day (Experimental): Participants received 30 mcg/kg/day serelaxin as continuous i.v. infusion for 48 hours.
  Interventions: Drug: Serelaxin
- Placebo (Placebo Comparator): Participants received continuous i.v. infusion of placebo matched to serelaxin for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serelaxin — Intravenous infusion
  Arms: Serelaxin 10 mcg/kg/Day; Serelaxin 30 mcg/kg/Day
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to assess safety, tolerability and pharmacokinetics and to explore efficacy of IV infusion of 10 µg/kg/day and 30 µg/kg/day serelaxin for 48 hours compared to placebo, when added to the standard therapy, in approximately 45 Japanese AHF patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent must be obtained before any study-specific assessment is performed.
* Male or female ≥20 years of age, with body weight ≥30 kg and ≤160 kg
* Hospitalized for AHF; AHF is defined as including all of the followings measured at any time between presentation (including the emergency department) and the end of screening:
* Dyspnea at rest or with minimal exertion
* Pulmonary congestion on chest radiograph
* BNP ≥350 pg/mL or NT-proBNP ≥1,400 pg/mL
* SBP ≥125 mmHg at the start and at the end of screening
* Able to be randomized within 16 hours from presentation to the hospital, including the emergency department
* Received intravenous (IV) furosemide of at least 40 mg (or equivalent) at any time between presentation (this include outpatient clinic, ambulance, or hospital including emergency department) and the start of screening for the study for the treatment of the current acute heart failure (HF) episode.
* Impaired renal function defined as an estimated glomerular filtration rate (eGFR) between presentation and randomization of ≥ 25 and≤ 75 mL/min/1.73 m2, calculated using the Japanese formula

Key Exclusion Criteria:

* Dyspnea primarily due to non-cardiac causes
* Temperature >38.5°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment
* Clinical evidence of acute coronary syndrome currently or within 30 days prior to enrollment.
* AHF due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate <45 beats per minute, or atrial fibrillation/flutter with sustained ventricular response of >130 beats per minute.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Japan (15):
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Ueda, Nagano
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Komatsushimachō, Tokushima
  - Novartis Investigative Site, Itabashi-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 centers in Japan.
Groups:
- Serelaxin 10 mcg/kg/Day: Participants received 10 micrograms/kilogram/day (mcg/kg/day) serelaxin as continuous intravenous (i.v.) infusion for 48 hours.
Period: Overall Study
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Started | 16 | 15 | 15
Completed | 16 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed on safety population defined as all randomized participants received any amount of study drug and had at least one post-baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (11.77) | 79.7 (9.01) | 76.4 (12.08) | 75.3 (11.54)
Age, Customized [Number; unit: participants]
  < 65 years | 6 | 1 | 3 | 10
  ≥ 65 years | 10 | 14 | 12 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 12
  Male | 12 | 10 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuations Due to AEs and SAEs, AEs Requiring Dose Adjustment or Interruption and Additional Therapy
Description: AEs were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. SAEs were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards. AEs leading to discontinuations, or requiring dose adjustment or interruptions and additional therapy were assessed.
Time Frame: From start of study treatment up to Day 5 (for AEs); From start of study treatment up to Day 14 (for SAEs)
Population: The analysis was performed on the safety population, defined as all participants who received at least one dose of study treatment and had at least one post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
participants
  AEs | 10 | 11 | 9
  SAEs | 1 | 3 | 0
  Death | 0 | 0 | 0
  Discontinuation due to AE(s) | 0 | 2 | 0
  Discontinuation due to SAE(s) | 0 | 0 | 0
  AEs requiring dose adjustment or interruption | 0 | 1 | 0
  AEs requiring additional therapy | 8 | 10 | 9
  AEs related to study drug | 2 | 2 | 0

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Serelaxin
Description: Maximum plasma concentration (Cmax) was defined as the peak level of serelaxin, derived from plasma concentration-time data, using a non-compartmental model approach.
Time Frame: Baseline (pre-dose), 1, 2, 24, 48, 49, 52 and 56 hours (post-dose)
Population: The analysis was performed in the pharmacokinetic (PK) set, defined as all participants who received study treatment and had at least one evaluable PK parameter data. Here, "Number of participants analyzed" signifies participants evaluable for this PK parameter at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram(s)/milliliter (ng/mL)
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day
Number analyzed (Participants) | 12 | 8
nanogram(s)/milliliter (ng/mL) | 8.01 (2.07) | 19.2 (4.69)

3. Primary Outcome: Weight Adjusted Clearance (CL) of Serelaxin
Description: Weight adjusted clearance (CL) was defined as the total body clearance of serelaxin after drug administration. CL was calculated as nominal infusion rate divided by Css, using a non-compartmental model approach.
Time Frame: Baseline (pre-dose), 1, 2, 24, 48, 49, 52 and 56 hours (post-dose)
Population: The analysis was performed in the PK population. Here, "Number of participants analyzed" signifies participants evaluable for this PK parameter at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day
Number analyzed (Participants) | 12 | 8
mL/hr/kg | 56.8 (15.4) | 70.2 (23.2)

4. Primary Outcome: Concentration at Steady-state (Css) of Serelaxin
Description: Concentration at steady-state (Css) was defined as concentration at the state of equilibrium obtained at the end of a certain number of administrations. Css of serelaxin in plasma was calculated by using a non-compartmental model approach.
Time Frame: Baseline (pre-dose), 1, 2, 24, 48, 49, 52 and 56 hours (post-dose)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day
Number analyzed (Participants) | 12 | 8
ng/mL | 7.81 (1.96) | 19.1 (4.61)

5. Secondary Outcome: Change From Baseline in Area Under the Curve (AUC) for Systolic Blood Pressure (SBP) Through 48 Hours of Infusion at Day 5
Description: The area under the curve (AUC) was defined as area under the plasma concentration-time curve from time zero to time of the last time point with measurable concentration, calculated by a trapezoidal method. Systolic blood pressure was measured using a calibrated standard sphygmomanometer after the subject remained in sitting position for 3 minutes at clinic during the visit. Sample collected at: Baseline; 30 & 60 minutes and then every hour for the first 6 hours of study drug infusion, and then every 3 hours during 48 hours of study drug infusion; every 3 hours until 12 hours following end of infusion, then every 6 hours for 48 hours and then every 24 hours until the earlier of Day 5 or discharge.
  AUC for SBP is standardized by dividing by the length of respective time ranges.
Time Frame: Baseline, 48 hours, Day 5
Population: The analysis was performed in the full analysis set (FAS) population, defined as all participants who were randomized in the study.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
mmHg
  48 hours | -8.21 (2.903) | -18.6 (3.018) | -10.88 (3.018)
  Day 5 | -8.79 (2.761) | -22.14 (2.871) | -14.77 (2.871)

6. Secondary Outcome: Change From Baseline in Aldosterone Levels Through Day 14
Description: Aldosterone biomarker was used to assess the effect of serelaxinin on fluid retention. Geometric means of the ratio of post-Baseline values to baseline values of aldosterone was calculated by treatment for the full analysis set.
Time Frame: Baseline, Day 1, Day 2, Day 5, Day 14
Population: The analysis was performed in the FAS population. Only participants with a value at both baseline and the post-dose time point were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Ratio
  Day 1 | 0.985 [0.7636 to 1.2717] | 0.816 [0.6118 to 1.0897] | 0.791 [0.6374 to 0.9825]
  Day 2 | 0.975 [0.7492 to 1.2685] | 0.721 [0.5195 to 0.9999] | 0.911 [0.7141 to 1.1620]
  Day 5 | 0.895 [0.6327 to 1.2656] | 0.825 [0.6468 to 1.0531] | 0.816 [0.5352 to 1.2452]
  Day 14 | 1.510 [0.9934 to 2.2962] | 1.114 [0.7983 to 1.5555] | 1.179 [0.8337 to 1.6661]

7. Secondary Outcome: Change From Baseline in Cystatin-C Levels Through Day 14
Description: Cystatin-C biomarker was used to assess the effect of serelaxinin on worsening of renal function. Geometric means of the ratio of post-Baseline values to baseline values of Cystatin-C was calculated by treatment for the full analysis set.
Time Frame: Baseline, Day 1, Day 2, Day 5, Day 14
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Ratio
  Day 1 | 0.921 [0.8863 to 0.9565] | 0.988 [0.9213 to 1.0598] | 0.985 [0.9291 to 1.0450]
  Day 2 | 0.930 [0.8736 to 0.9900] | 0.852 [0.6465 to 1.1236] | 0.965 [0.9002 to 1.0346]
  Day 5 | 1.062 [0.9898 to 1.1384] | 1.115 [1.0207 to 1.2178] | 1.038 [0.9627 to 1.1194]
  Day 14 | 1.195 [1.0154 to 1.4057] | 1.136 [1.0348 to 1.2472] | 1.125 [1.0313 to 1.2271]

8. Secondary Outcome: Change From Baseline in High Sensitivity Troponin-T Levels Through Day 14
Description: High sensitivity Troponin-T biomarker was used to assess the effect of serelaxin on myocardial damage. Geometric means of the ratio of post-Baseline values to baseline values of high sensitivity troponin-t was calculated by treatment for the full analysis set.
Time Frame: Baseline, Day 1, Day 2, Day 5, Day 14
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Ratio
  Day 1 | 0.899 [0.7598 to 1.0643] | 1.060 [0.8932 to 1.2572] | 0.956 [0.8652 to 1.0559]
  Day 2 | 0.856 [0.6935 to 1.0553] | 1.040 [0.8514 to 1.2714] | 0.894 [0.7650 to 1.0442]
  Day 5 | 0.849 [0.5984 to 1.2044] | 0.972 [0.7779 to 1.2151] | 0.779 [0.5250 to 1.1572]
  Day 14 | 0.820 [0.5729 to 1.1730] | 0.813 [0.4480 to 1.4748] | 0.685 [0.4652 to 1.0093]

9. Secondary Outcome: Change From Baseline in NT-proBNP Levels Through Day 14
Description: NT-proBNP biomarker was used to assess the effect of serelaxinin on degree of cardiac wall stress and congestion. Geometric means of the ratio of post-Baseline values to baseline values of NT-proBNP was calculated by treatment for the full analysis set.
Time Frame: Baseline, Day 1, Day 2, Day 5, Day 14
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Ratio
  Day 1 | 0.585 [0.4356 to 0.7865] | 0.646 [0.5146 to 0.8115] | 0.673 [0.5416 to 0.8363]
  Day 2 | 0.492 [0.3421 to 0.7076] | 0.451 [0.3271 to 0.6210] | 0.581 [0.4410 to 0.7656]
  Day 5 | 0.388 [0.2502 to 0.6028] | 0.386 [0.2575 to 0.5796] | 0.526 [0.3685 to 0.7503]
  Day 14 | 0.295 [0.1649 to 0.5293] | 0.419 [0.2621 to 0.6691] | 0.277 [0.1875 to 0.4079]

10. Secondary Outcome: Change From Baseline in Neutrophil Gelatinase-asc Lipocalin (NGAL) Levels Through Day 14
Description: Neutrophil gelatinase-asc lipocalin (NGAL) biomarker was used to assess the effect of serelaxin on kidney function. Geometric means of the ratio of post-Baseline values to baseline values of NGAL was calculated by treatment for the full analysis set.
Time Frame: Baseline, Day 1, Day 2, Day 5, Day 14
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Number analyzed (Participants) | 16 | 15 | 15
Ratio
  Day 1 | 1.011 [0.8911 to 1.1478] | 1.083 [0.9025 to 1.2996] | 1.054 [0.9574 to 1.1613]
  Day 2 | 0.929 [0.8443 to 1.0229] | 1.172 [0.9994 to 1.3736] | 1.099 [0.9866 to 1.2236]
  Day 5 | 1.129 [1.0145 to 1.2560] | 1.238 [1.0139 to 1.5114] | 1.135 [1.0141 to 1.2698]
  Day 14 | 1.434 [1.1760 to 1.7489] | 1.520 [1.3214 to 1.7485] | 1.433 [1.1793 to 1.7401]

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit
Arm/Group | Serelaxin 10 mcg/kg/Day | Serelaxin 30 mcg/kg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/16 | 3/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/16 | 9/15 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin 10 mcg/kg/Day (N=16) | Serelaxin 30 mcg/kg/Day (N=15) | Placebo (N=15)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin 10 mcg/kg/Day (N=16) | Serelaxin 30 mcg/kg/Day (N=15) | Placebo (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 4 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
INFUSION SITE PAIN (General disorders) | 1 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0 | 0
BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0
BLOOD PRESSURE DECREASED (Investigations) | 1 | 1 | 0
BLOOD PRESSURE SYSTOLIC DECREASED (Investigations) | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0
DELIRIUM (Psychiatric disorders) | 1 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1
RESTLESSNESS (Psychiatric disorders) | 1 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1 | 0
GENITAL PAIN (Reproductive system and breast disorders) | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
VASCULITIS (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single--site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.